CLINICAL TRIAL: NCT05773599
Title: The Evaluation of the Effect of Laughter Yoga on Sleep Quality and Life Satisfaction in Midwifery Students
Brief Title: Midwifery Students and Laughter Yoga
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Safiye AĞAPINAR ŞAHİN, Asst. Prof., Ataturk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Ataturk University SSAHIN0001
Record Dates: First submitted 2023-01-23; First posted 2023-03-17 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Laughter Yoga; Midwifery; Life Satisfaction
Keywords: Yoga; Laughter; student; sleep; life
MeSH Terms: conditions — Personal Satisfaction; Laughter | interventions — Laughter Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- laughter yoga (Experimental): A pre-test will be applied to evaluate sleep quality and life satisfaction. 4 sessions of laughter yoga will be applied to the experimental group with a low sleep quality score, one day apart. Afterwards, sleep quality and life satisfaction will be evaluated with the posttest.
  Interventions: Other: laughter yoga
- kontrol (No Intervention): A pre-test will be applied to evaluate sleep quality and life satisfaction. The control group with a low sleep quality score will not receive any intervention. In parallel with the experimental group, sleep quality and life satisfaction will be evaluated again with the posttest.

INTERVENTIONS:
Other: laughter yoga — A pre-test will be applied to evaluate sleep quality and life satisfaction. Laughter yoga will be applied one day apart to the experimental group with a low sleep quality score. After dasa, sleep quality and life satisfaction will be evaluated again with
  Arms: laughter yoga

SUMMARY:
No study was found as a result of the literature review. It is thought that laughter yoga will affect the life satisfaction and sleep quality of individuals due to reasons such as increasing oxygen saturation in the blood, strengthening mental functions, providing mental well-being and reducing stress. stress and mental fatigue are thought to affect life satisfaction and sleep quality, so it was planned to evaluate the effect of laughter yoga on life satisfaction and sleep quality.

DETAILED DESCRIPTION:
With laughter, oxygen saturation in the brain and body increases. Laughter yoga basically includes breathing, meditation and different stretching movements. Benefits of laughter yoga; relaxes the muscles, reduces the level of stress hormones, ensures effective breathing, increases pain tolerance, strengthens mental functions, stimulates the circulatory and immune system, reduces anxiety and depression symptoms, improves quality of life and creates psychosocial well-being. Life satisfaction is the result obtained by comparing the expectations of the individual with what he has. Life satisfaction is affected by many factors such as daily stress, work life, social relations, and mental state. Life satisfaction is not related to certain areas, but to be happy in all areas of life.

Sleep is of great importance in fulfilling daily functions and in maintaining mental and physical health. sleep quality; It is the quantitative evaluation of sleep such as the time to fall asleep, the total time spent in sleep, the number of awakenings, and the duration of awakening.

ELIGIBILITY:
Inclusion Criteria:

* Students who agreed to participate in the study

Exclusion Criteria:

* not be a midwifery student

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2023-01-13 (Actual); Study Completion 2023-01-27 (Actual)

PRIMARY OUTCOMES:
The effect of laughter yoga on life satisfaction | one day
  The life satisfaction of students will be measured with the life satisfaction scale. The "Satisfaction with Life Scale", whose validity and reliability study was conducted in Turkish by Dağlı and Baysal in 2016, has a total of five items and a 5-point Likert type, and the internal consistency coefficient of the scale has been reported to be 0.92. A high score from the scale, which has a single factor structure, indicates that the individual's life satisfaction is high.
The effect of laughter yoga on sleep quality | 28 day
  The Cronbach's alpha internal consistency coefficient of the original scale was calculated as 0.83 and the Turkish version was 0.80. PUKI consists of 24 questions in total. The last 5 questions on the scale must be answered by the spouse or roommate. These 5 questions are used for clinical information only and are not included in the scoring. Therefore, 18 items are included in the scoring in PUKI. The questions consist of seven sub-components: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, use of sleep medication, and daytime dysfunction. Each question is evaluated by giving points between 0-3. The sum of the scores of these seven sub-components constitutes the total score of PUKI. The total PUKI score has a value between 0-21. Sleep quality of those with a total score of 5 and less than 5 was "good"; Sleep quality of those with a score greater than 5 is considered "poor".

CONTACTS AND LOCATIONS:
Overall Officials: Safiye Ağapınar Şahin, Ass.Dr., Principal Investigator — Atatürk University Faculty of Health Sciences Department of Midwifery Yakutiye/Erzurum; Sibel Öztürk, Ass. Dr., Study Director — Atatürk University Faculty of Health Sciences Department of Midwifery Yakutiye/Erzurum; Nazlı Akar, assistant, Study Director — research assistant
Locations (1):
- Atatürk University Faculty of Health Sciences Department, Erzurum, Yakuti̇ye/erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
We do not share Individual Participant data with other researchers.